CLINICAL TRIAL: NCT04378634
Title: The Influence of Epigenetic Modifications and Post-Exertional Malaise in People With Myalgic Encephalomyelitis/Chronic Fatigue Syndrome
Brief Title: Epigenetics of Post-exertional Malaise in Patients With ME/CFS
Acronym: EPIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Andrea Polli, PhD, principal investigator, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EPIME
Record Dates: First submitted 2020-04-27; First posted 2020-05-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Fatigue Syndrome, Chronic
Keywords: Chronic Fatigue Syndrome; Exercise; Epigenetics; DNA methylation
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ME/CFS Exercise (Experimental): Patients undergoing the physical stress test (aerobic power index)
  Interventions: Behavioral: Exercise; Other: Mental Stress Test
- Patients Stress (Experimental): Patients undergoing the mental stress task (MIST)
  Interventions: Behavioral: Exercise; Other: Mental Stress Test
- Healthy Exercise (Active Comparator): Healthy controls undergoing the physical stress test (aerobic power index)
  Interventions: Behavioral: Exercise; Other: Mental Stress Test
- Healthy Stress (Active Comparator): Healthy controls undergoing the mental stress task (MIST)
  Interventions: Behavioral: Exercise; Other: Mental Stress Test

INTERVENTIONS:
Behavioral: Exercise — Sub-maximal exercise test
  Other Names: Aerobic Power Index
Other: Mental Stress Test — Computerised mental arithmetic challenges and social evaluative threat tasks
  Other Names: Montreal Imaging Stress Task

SUMMARY:
Exploring epigenetic mechanisms of Myalgic Encephalomyelitis / Chronic Fatigue Syndrome (ME/CFS) is crucial to understand the mechanisms underlying its pathophysiology. Three potential candidates have been selected (BDNF, COMT, and HDAC genes). DNA methylation in the promoter regions of those genes will be explored.

The investigators designed a randomised controlled trial and will enrol 70 patients with ME/CFS and 35 age-, sex-, and BMI-matched healthy controls. Both groups will be randomised in 2 groups and receive either one session of aerobic exercise or a validated test designed to trigger mental stress and mental fatigue. The primary aim is to assess genetic and epigenetic mechanisms of BDNF, COMT and HDAC genes in response to exercise and the stress task.

DETAILED DESCRIPTION:
The only way to improve the diagnosis and treatment of Myalgic Encephalomyelitis / Chronic Fatigue Syndrome (ME/CFS) is to better understand the mechanisms underlying its pathophysiology. Central nervous system dysfunctions play a major role in ME/CFS and help explaining patients' symptoms, such as general malaise occurring after physical activity (i.e. post-exertional malaise). Therefore, post-exertional malaise in relation to three major candidates involved in central nervous system functioning - brain-derived neurotrophic factor (BDNF), catechol-O-methyltransferase (COMT) and histone de-acetylases (HDAC) - will be explored.

BDNF is a protein involved in crucial functions such as nerve growth, memory and learning, and plays a role in neuronal sensitisation and pain. However, no study has explored the role of BDNF in ME/CFS. Our research group performed a preliminary study which focussed on BDNF in ME/CFS. In a previous study, the investigators assessed DNA methylation (an epigenetic mechanism that contribute to gene expression silencing), and protein expression in serum of the BDNF in patients with ME/CFS and healthy controls. Patients showed significantly less DNA methylation and significantly more BDNF protein. Given these exciting findings, further study is warranted.

COMT is an enzyme encoded by its homonymous gene. The enzyme degrades catecholamines like dopamine, epinephrine and norepinephrine. Catecholamines have been repeatedly associated with pain, stress, and depression. Lower COMT activity increases catecholamines level, causes hyperalgesia, and has been associated with depressive symptoms.

Similarly, research on histone acetylation shows that another group of enzymes (Histone de-acetylases, HDACs) are increased during neural sensitisation and pain. However, no research has been done on HDACs in patients with ME/CFS. Interestingly, aerobic exercise has been shown to increase BDNF release and decrease COMT and HDACs activity. Given the detrimental acute effects that exercise can have on patients with ME/CFS, investigators hypothesised that understanding the role of BDNF, COMT, and HDACs following exercise would help elucidating both mechanisms of post-exertional malaise and ME/CFS pathophysiology.

A randomised controlled trial has been designed including 70 patients with ME/CFS and 35 age-, sex-, and BMI-matched healthy controls. Both groups will be randomised in 2 groups. One group will undergo one session of aerobic exercise, and the other group undergoes a validated test designed to trigger mental stress and mental fatigue. All participants will undergo clinical assessments, measurements of pain thresholds, and blood withdrawal before and after the exercise/mental stress exposure. The aims are to assess genetic and epigenetic mechanisms of BDNF, COMT and HDAC genes, as well as the expression of these factors in blood and serum in patients with ME/CFS.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ME/CFS established by a MD experienced in the field of internal medicine and ME/CFS - according to the published international criteria developed by the Canadian Consensus Criteria (CCC);
* age between 18 and 70 years old;
* body mass index (BMI) below 30 (no obesity).

Exclusion Criteria:

* presence of other neurological disorders (Parkinson's disease, Multiple Sclerosis, etc);
* presence of systemic disorders (lupus erythematosus, rheumatoid arthritis, etc.);
* presence or history of cardiac disorders (coronary heart disease, history of heart failure, etc);
* presence or history of cancer;
* presence or history of neuropathic pain (e.g. pain related to herpes zoster virus);
* pregnancy;

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
DNA methylation | Baseline through 1 week post intervention
  DNA methylation measured at several CpGs of the genes' promoter regions using pyrosequencing technology

SECONDARY OUTCOMES:
Clinical Symptoms | Baseline through 1 week post intervention
  Symptoms reported by the patients using the DePaul Symptoms Questionniare
Pain sensitivity | Baseline through 1 week post intervention
  Sensitivity to mechanical stimuli using a digital algometer (FPXTM, Fisher, Wagner Instruments, Greenwich) as well as heat and cold stimuli using the TSA-II device (Medoc, CA, USA). The devices will be placed, in random order to prevent test order effects, at three different body sites: the skin web between thumb and index finger, trapezius muscle, and proximal third of tibialis anterior muscle, in order to test pain thresholds on non-specific locations both on the extremities and the trunk.
Serum BDNF | Baseline through 1 week post intervention
  BDNF protein expression in serum using Enzyme-Linked Immunosorbent Assay (ELISA) kit for human BDNF
Cortisol response | Baseline through 1 week post intervention
  Cortisol will be measured in saliva and used as a measure of stress responses using LC/MS-MS method.

OTHER OUTCOMES:
General Health | Baseline
  General health will be measured using the Short Form-36 Health Survey (SF-36) questionnaire. The questionnaire returns a score from 0 to 100 where higher scores mean less disability.
Gene's polymorphisms | Baseline
  Genes' polymorphisms might mediate epigenetic changes. They will be assessed using pyrosequencing technology.

CONTACTS AND LOCATIONS:
Overall Officials: Jo Nijs, PhD, Study Director — Vrije Universiteit Brussel
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Vega WC, Vernon SD, McGowan PO. DNA methylation modifications associated with chronic fatigue syndrome. PLoS One. 2014 Aug 11;9(8):e104757. doi: 10.1371/journal.pone.0104757. eCollection 2014. PMID 25111603
- [Background] Vangeel EB, Kempke S, Bakusic J, Godderis L, Luyten P, Van Heddegem L, Compernolle V, Persoons P, Lambrechts D, Izzi B, Freson K, Claes S. Glucocorticoid receptor DNA methylation and childhood trauma in chronic fatigue syndrome patients. J Psychosom Res. 2018 Jan;104:55-60. doi: 10.1016/j.jpsychores.2017.11.011. Epub 2017 Nov 20. PMID 29275786
- [Background] Trivedi MS, Oltra E, Sarria L, Rose N, Beljanski V, Fletcher MA, Klimas NG, Nathanson L. Identification of Myalgic Encephalomyelitis/Chronic Fatigue Syndrome-associated DNA methylation patterns. PLoS One. 2018 Jul 23;13(7):e0201066. doi: 10.1371/journal.pone.0201066. eCollection 2018. PMID 30036399